CLINICAL TRIAL: NCT04067076
Title: Massive Mental Health Screening Using Smartphones in 24 Pre-graduate Education Centers in Mexico City: TEDUCA Survey Protocol
Acronym: TEDUCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); Instituciones Educativas de nivel Medio Superior (IEMS) de Ciudad de México (Unknown); Gobierno de la Ciudad de Mexico (Unknown)
Responsible Party: Sponsor
Other Study IDs: SmartMexSurvey2
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Suicidal Ideation; Social Behavior; Depression; Depressive Disorder; Anxiety; Alcohol Drinking; Drug Abuse
Keywords: Mass Screening; Health Surveys; Mental Health; Suicidal Ideation; Young Adult; Interpersonal Relations; Smartphone
MeSH Terms: conditions — Suicidal Ideation; Social Behavior; Depression; Depressive Disorder; Anxiety Disorders; Alcohol Drinking; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students of IEMS of Mexico City: Students currently enrolled in the academic year 2019-2020 from the 24 IEMS centers of Mexico City
  Interventions: Other: Self-administered evaluation questionnaire

INTERVENTIONS:
Other: Self-administered evaluation questionnaire — Smartphone app with MeMind questionnaires

SUMMARY:
The objective of this study is to make a massive suicide risk and social behavior assessment in 24 pre-graduate education centers in Mexico City (approximately 30,000 students aged between 15 and 22 years), taking also into account other outcomes such as depression, anxiety, alcohol and drugs. For this, an app for Smartphone (MeMind) or a web platform (www.MeMind.net) will be used in which the participants will take a self-administered questionnaire, composed of several psychometric instruments.

Our main hypothesis is that identification of suicide risk in the Mexico City's student community is feasible using their own smartphones and can serve as both a population screening tool for early specialist referral, as well as a tool for evaluating social behavior strategies and their relation to suicide behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Use a smartphone as personal or computer terminals enabled by the municipality of Milpa Alta or educational services.
2. Be able to understand the nature, purpose and methodology of the study.
3. Accept participation in the study and check the corresponding box in the app to verify that the informed consent has been expressly given.

Exclusion Criteria:

1. Subject deprived of liberty (by judicial or administrative decision)
2. Subject protected by law (guardianship or conservatorship)

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community composed of students between 15 and 22 years of the 24 educational institutions IEMS of Mexico City, enrolled at the scholar year 2019-2020
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation | 1 Day
  Columbia-Suicide Severity Rating Scale (C-SSRS) is encompassed into MeMind for this purpose.
  In C-SSRS, four constructs are measured. The first is the severity of ideation, which is rated on a 5-point ordinal scale from 1="wish to be dead" to 5="suicidal intent with plan".
  The second is the intensity of ideation, which comprises 5 items, each rated on a 5-point ordinal scale: frequency, duration, controllability, deterrents, and reason for ideation.
  The third is the behavior, which is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
  And the fourth is the lethality, which assesses actual attempts; actual lethality is rated on a 6-point ordinal scale.
  Results are coded in the instrument itself with colored labels that indicates definitions of suicidal ideation and behavior, quantify both of them and gauge their severity.
  Definitions are available elsewhere (http://cssrs.columbia.edu).
Social Behavior | 1 Day
  The assessment of social interaction will be carried out through six games that expose the participant to decision-making in preset environments with very simple and easily understandable rules (Dictator's Game, Prisoner's Dilemma, Loss Aversion, Risk Aversion, Trust Game or The Investment Game, and Ambiguity Aversion).

SECONDARY OUTCOMES:
Depression | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to depression.
  PHQ-9 questionnaire is emcompassed into Memind for this purpose.
Anxiety | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to anxiety.
  GAD-7 (only screeni
Drug Utilization | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to drug abuse.
  DAST (only questions 1,6,7) is emcompassed into Memind for this purpose.
Alcohol Drinking | 1 Day
  Participants will be asked to complete a questionnaire regarding possible symptoms related to alcohol abuse.
  Alcohol Use Disorders Identification Test (AUDIT-C)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcaldía Milpa Alta. Ciudad de México, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for researchers upon request
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Upon request to Enrique Baca Garcia (enrique.baca@uam.es)

REFERENCES:
- [Derived] Martinez-Nicolas I, Arenas Castaneda PE, Molina-Pizarro CA, Rosado Franco A, Maya-Hernandez C, Barahona I, Martinez-Ales G, Aroca Bisquert F, Baca-Garcia E, Barrigon ML. Impact of Depression on Anxiety, Well-being, and Suicidality in Mexican Adolescent and Young Adult Students From Mexico City: A Mental Health Screening Using Smartphones. J Clin Psychiatry. 2022 Apr 6;83(3):20m13806. doi: 10.4088/JCP.20m13806. PMID 35390233
- See also: Related Info — http://www.MeMind.net